CLINICAL TRIAL: NCT00575744
Title: Sentinel Lymph Node Biopsy Using Peritumoral Injection With Blue Dye Confirmation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UAMS 04959
Record Dates: First submitted 2007-12-14; First posted 2007-12-18 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Breast Cancer
Keywords: Sentinel Lymph Node Biopsy; Axillary Node Dissection; Intraoperative Injection; Lumpectomy; Mastectomy
MeSH Terms: conditions — Breast Neoplasms | interventions — Sentinel Lymph Node Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (No Intervention)
  Interventions: Procedure: Sentinel Node Biopsy

INTERVENTIONS:
Procedure: Sentinel Node Biopsy — Once the patient is asleep under anesthetic, they receive an intraoperative injection of 1.0 mCi of Technetium-99 sulfur colloid into normal breast tissue surrounding the primary cancer or biopsy cavity directed subareolar or around the tumor. This is followed by blue dye injected in the subareolar complex approximately 5 minutes prior to incision. The sentinel node biopsy is performed, followed by lumpectomy/mastectomy, and a completion axillary node dissection if the sentinel node(s) were positive.
  Other Names: Axillary Node Dissection; Technitium Sulfur Colloid; Lymphazurin Blue Dye

SUMMARY:
We continue to collect information in support of the hypothesis that the histology of the first draining lymph node (sentinel node) accurately predicts the histology of the rest of the axillary lymph nodes.

DETAILED DESCRIPTION:
Using a technique combining Technetium-99 sulfur colloid and Lymphazurin Blue Dye, we have established that the sentinel node predicts the pathology results of the rest of the axillary lymph nodes. This minimally invasive technique, which can be readily performed under local anesthesia, makes the need for full axillary lymph node dissection unnecessary for most patients. If the sentinel node is negative, no further surgery is necessary. If positive, a complete axillary node dissection is performed. In addition, the injections are made while the patient is under anesthesia, reducing the physical and psychological pain that accompanies injections done pre-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer requiring lymph node evaluation
* Clinically negative lymph nodes in the axilla
* Willing participation following an informed consent process

Exclusion Criteria:

* Patients with clinically positive lymph nodes
* Pregnancy (if a pregnant female should be diagnosed with breast cancer an exception would be considered on a case to case basis)
* Previous axillary lymphadenectomy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 699 (Actual)
Dates: Start 1998-12; Primary Completion 2010-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
To continue gathering data relating to the sentinel lymph node biopsy procedure. | Time of surgery and data analysis

SECONDARY OUTCOMES:
To vary the techniques used in the multicenter trial and incorporate the use of blue dye along with the Technetium-99 sulfur colloid. | Time of surgery and data analysis

CONTACTS AND LOCATIONS:
Overall Officials: V. Suzanne Klimberg, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas For Medical Sciences, Little Rock, Arkansas, United States

REFERENCES:
- [Background] Layeeque R, Henry-Tillman R, Korourian S, Kass R, Klimberg VS. Subareolar sentinel node biopsy for multiple breast cancers. Am J Surg. 2003 Dec;186(6):730-5; discussion 735-6. doi: 10.1016/j.amjsurg.2003.08.014. PMID 14672787
- [Background] Rubio IT, Klimberg VS. Techniques of sentinel lymph node biopsy. Semin Surg Oncol. 2001 Apr-May;20(3):214-23. doi: 10.1002/ssu.1036. PMID 11523106
- [Background] Smith LF, Cross MJ, Klimberg VS. Subareolar injection is a better technique for sentinel lymph node biopsy. Am J Surg. 2000 Dec;180(6):434-7; discussion 437-8. doi: 10.1016/s0002-9610(00)00521-3. PMID 11182393
- [Background] Smith LF, Rubio IT, Henry-Tillman R, Korourian S, Klimberg VS. Intraoperative ultrasound-guided breast biopsy. Am J Surg. 2000 Dec;180(6):419-23. doi: 10.1016/s0002-9610(00)00500-6. PMID 11182390
- [Background] Klimberg VS, Rubio IT, Henry R, Cowan C, Colvert M, Korourian S. Subareolar versus peritumoral injection for location of the sentinel lymph node. Ann Surg. 1999 Jun;229(6):860-4; discussion 864-5. doi: 10.1097/00000658-199906000-00013. PMID 10363900
- [Background] McMasters KM, Giuliano AE, Ross MI, Reintgen DS, Hunt KK, Byrd DR, Klimberg VS, Whitworth PW, Tafra LC, Edwards MJ. Sentinel-lymph-node biopsy for breast cancer--not yet the standard of care. N Engl J Med. 1998 Oct 1;339(14):990-5. doi: 10.1056/NEJM199810013391410. No abstract available. PMID 9753717
- [Background] Krag D, Weaver D, Ashikaga T, Moffat F, Klimberg VS, Shriver C, Feldman S, Kusminsky R, Gadd M, Kuhn J, Harlow S, Beitsch P. The sentinel node in breast cancer--a multicenter validation study. N Engl J Med. 1998 Oct 1;339(14):941-6. doi: 10.1056/NEJM199810013391401. PMID 9753708
- [Result] Layeeque R, Kepple J, Henry-Tillman RS, Adkins L, Kass R, Colvert M, Gibson R, Mancino A, Korourian S, Klimberg VS. Intraoperative subareolar radioisotope injection for immediate sentinel lymph node biopsy. Ann Surg. 2004 Jun;239(6):841-5; discussion 845-8. doi: 10.1097/01.sla.0000128304.13522.00. PMID 15166963
- [Result] Thompson M, Korourian S, Henry-Tillman R, Adkins L, Mumford S, Smith M, Klimberg VS. Intraoperative radioisotope injection for sentinel lymph node biopsy. Ann Surg Oncol. 2008 Nov;15(11):3216-21. doi: 10.1245/s10434-008-0010-3. Epub 2008 Sep 6. PMID 18777194
- [Result] Johnson CB, Boneti C, Korourian S, Adkins L, Klimberg VS. Intraoperative injection of subareolar or dermal radioisotope results in predictable identification of sentinel lymph nodes in breast cancer. Ann Surg. 2011 Oct;254(4):612-8. doi: 10.1097/SLA.0b013e31823005bf. PMID 21918427